CLINICAL TRIAL: NCT03826927
Title: New Oral Anticoagulants in Stroke Patients-Long Term Prevention of Recurrent Stroke in Patients With Atrial Fibrillation- a National Prospective Registry (NOACISP Long Term)
Brief Title: New Oral Anticoagulants (NOAC) in Stroke Patients
Acronym: NOACISPLongTer
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: PB_2016-00662; me14Engelter2
Record Dates: First submitted 2019-01-22; First posted 2019-02-01 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Stroke; Atrial Fibrillation
Keywords: New oral Anticoagulants (NOAC); vitamin K antagonists (VKA); cerebrovascular disease
MeSH Terms: conditions — Stroke; Atrial Fibrillation; Cerebrovascular Disorders | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AF and cerebrovascular event: patients with AF and recent (< 3 month) stroke or transient ischaemic attack (TIA) or intracranial haemorrhage (ICH) with or without pre-existing oral anticoagulation, in whom treatment with NOACs or VKAs is initiated or continued for prevention of ischemic events
  Interventions: Other: treatment with NOACs or VKAs

INTERVENTIONS:
Other: treatment with NOACs or VKAs — treatment with NOACs or VKAs initiated or continued for prevention of ischemic events

SUMMARY:
Registry to explore characteristics, use and management of new oral anticoagulants (NOAC) and vitamin K antagonists (VKA) treatment among patients with atrial fibrillation (AF) and recent cerebrovascular disease in a "real-world" setting at a stroke centre.

DETAILED DESCRIPTION:
Registry to explore characteristics, use and management of new oral anticoagulants (NOAC) and vitamin K antagonists (VKA) treatment among patients with atrial fibrillation (AF) and recent cerebrovascular disease in a "real-world" setting at a stroke centre. Special interest is payed to conditions not or only in part investigated in the large randomised controlled Trials (RCT) and that are specific to patients with cerebrovascular disease. This includes early start of NOAC treatment after recent stroke, very old patients, multimorbidity, patients with a history of intracranial haemorrhage (ICH) and patient satisfaction and preferences with VKA/NOACS.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent form (ICF)
* existing or newly diagnosed AF
* recent (< 3 month) stroke (ischemic or haemorrhagic) or TIA (=index event)
* treatment with NOACs or VKAs is continued, changed or initiated for prevention of ischemic events

Exclusion Criteria:

* patients not able or unwilling to sign ICF
* patient is, in the opinion of the investigator, unlikely to comply with the scheduled follow-up visits or is unsuitable for any other reason
* patients who will not be anticoagulated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients eligible for this registry will be recruited at the stroke centre at the University Hospital Basel
Sampling Method: Probability Sample
Enrollment: 1023 (Actual)
Dates: Start 2013-03-01 (Actual); Primary Completion 2021-08 (Actual); Study Completion 2021-08 (Actual)

PRIMARY OUTCOMES:
Change in anticoagulation (NOAC and VKA) treatment | time from index event (= cerebrovascular event) to Follow- up assessments at 3-, 6-, 12- and 24 months after index event
  assessment of details of NOAC or VKA application (start, pause, dosage)

SECONDARY OUTCOMES:
Change in glomerular filtration rate (GFR) | time from index event (= cerebrovascular event) to Follow- up assessments at 3-, 6-, 12- and 24 months after index event
  impact of kidney function (in particular volatile GFR (ml/min) around the threshold for reduced dosage)
Drug adherence for anticoagulation (VKA) treatment | time from index event (= cerebrovascular event) to Follow- up assessments at 3-, 6-, 12- and 24 months after index event
  monitor the frequency of VKA use in patients with stroke or TIA attributable to AF, (a) among patients without pre-existing anticoagulation, (b) among patients under insufficient VKA therapy, and (c) among patients with sufficient VKA therapy, assessed by telephone or clinical visit
Change in anticoagulant treatment | time from index event (= cerebrovascular event) to Follow- up assessments at 3-, 6-, 12- and 24 months after index event
  If anticoagulant treatment was stopped or switched to any other drug (NOAC/VKA), reason for switching will be documented
Recording of Adverse Events (AE) | time from index event (= cerebrovascular event) to Follow- up assessments at 3-, 6-, 12- and 24 months after index event
  Causality for AE will be assessed as related, possibly related or non-related to the prescribed anticoagulant
Change in modified Rankin Scale (mRS) | time from index event (= cerebrovascular event) to Follow- up assessments at 3-, 6-, 12- and 24 months after index event
  modified Rankin Scale (mRS) is a scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability; scale runs from 0-6, running from perfect health (=0) without symptoms to death (=6)
Co-morbidities | time from index event (= cerebrovascular event) to Follow- up assessments at 3-, 6-, 12- and 24 months after index event
  Recording of co-morbidities
Drug adherence for anticoagulation (NOAC) treatment | time from index event (= cerebrovascular event) to Follow- up assessments at 3-, 6-, 12- and 24 months after index event
  monitor the frequency of NOAC use in patients with stroke or TIA attributable to AF, assessed by telephone or clinical visit

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Lyrer, Prof. Dr. MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (2):
- Switzerland (2):
  - Felix Platter Spital, Basel
  - Dep. of Neurology, Hospital of the University of Basel, Basel

REFERENCES:
- [Background] Polymeris AA, Zietz A, Schaub F, Meya L, Traenka C, Thilemann S, Wagner B, Hert L, Altersberger VL, Seiffge DJ, Lyrer F, Dittrich T, Piot I, Kaufmann J, Barone L, Dahlheim L, Flammer S, Avramiotis NS, Peters N, De Marchis GM, Bonati LH, Gensicke H, Engelter ST, Lyrer PA. Once versus twice daily direct oral anticoagulants in patients with recent stroke and atrial fibrillation. Eur Stroke J. 2022 Sep;7(3):221-229. doi: 10.1177/23969873221099477. Epub 2022 May 10. PMID 36082252
- [Background] Kimura S, Toyoda K, Yoshimura S, Minematsu K, Yasaka M, Paciaroni M, Werring DJ, Yamagami H, Nagao T, Yoshimura S, Polymeris A, Zietz A, Engelter ST, Kallmunzer B, Cappellari M, Chiba T, Yoshimoto T, Shiozawa M, Kitazono T, Koga M; SAMURAI, RELAXED, RAF, RAF-NOAC, CROMIS-2, NOACISP LONGTERM, Erlangen Registry and Verona Registry Investigators. Practical "1-2-3-4-Day" Rule for Starting Direct Oral Anticoagulants After Ischemic Stroke With Atrial Fibrillation: Combined Hospital-Based Cohort Study. Stroke. 2022 May;53(5):1540-1549. doi: 10.1161/STROKEAHA.121.036695. Epub 2022 Feb 2. PMID 35105180
- [Background] Seiffge DJ, De Marchis GM, Koga M, Paciaroni M, Wilson D, Cappellari M, Macha Md K, Tsivgoulis G, Ambler G, Arihiro S, Bonati LH, Bonetti B, Kallmunzer B, Muir KW, Bovi P, Gensicke H, Inoue M, Schwab S, Yaghi S, Brown MM, Lyrer P, Takagi M, Acciarrese M, Jager HR, Polymeris AA, Toyoda K, Venti M, Traenka C, Yamagami H, Alberti A, Yoshimura S, Caso V, Engelter ST, Werring DJ; RAF, RAF-DOAC, CROMIS-2, SAMURAI, NOACISP, Erlangen, and Verona registry collaborators. Ischemic Stroke despite Oral Anticoagulant Therapy in Patients with Atrial Fibrillation. Ann Neurol. 2020 Feb 12;87(5):677-87. doi: 10.1002/ana.25700. Online ahead of print. PMID 32052481
- [Background] Wilson D, Ambler G, Lee KJ, Lim JS, Shiozawa M, Koga M, Li L, Lovelock C, Chabriat H, Hennerici M, Wong YK, Mak HKF, Prats-Sanchez L, Martinez-Domeno A, Inamura S, Yoshifuji K, Arsava EM, Horstmann S, Purrucker J, Lam BYK, Wong A, Kim YD, Song TJ, Schrooten M, Lemmens R, Eppinger S, Gattringer T, Uysal E, Tanriverdi Z, Bornstein NM, Assayag EB, Hallevi H, Tanaka J, Hara H, Coutts SB, Hert L, Polymeris A, Seiffge DJ, Lyrer P, Algra A, Kappelle J, Al-Shahi Salman R, Jager HR, Lip GYH, Mattle HP, Panos LD, Mas JL, Legrand L, Karayiannis C, Phan T, Gunkel S, Christ N, Abrigo J, Leung T, Chu W, Chappell F, Makin S, Hayden D, Williams DJ, Kooi ME, van Dam-Nolen DHK, Barbato C, Browning S, Wiegertjes K, Tuladhar AM, Maaijwee N, Guevarra C, Yatawara C, Mendyk AM, Delmaire C, Kohler S, van Oostenbrugge R, Zhou Y, Xu C, Hilal S, Gyanwali B, Chen C, Lou M, Staals J, Bordet R, Kandiah N, de Leeuw FE, Simister R, van der Lugt A, Kelly PJ, Wardlaw JM, Soo Y, Fluri F, Srikanth V, Calvet D, Jung S, Kwa VIH, Engelter ST, Peters N, Smith EE, Yakushiji Y, Orken DN, Fazekas F, Thijs V, Heo JH, Mok V, Veltkamp R, Ay H, Imaizumi T, Gomez-Anson B, Lau KK, Jouvent E, Rothwell PM, Toyoda K, Bae HJ, Marti-Fabregas J, Werring DJ; Microbleeds International Collaborative Network. Cerebral microbleeds and stroke risk after ischaemic stroke or transient ischaemic attack: a pooled analysis of individual patient data from cohort studies. Lancet Neurol. 2019 Jul;18(7):653-665. doi: 10.1016/S1474-4422(19)30197-8. Epub 2019 May 23. PMID 31130428
- [Background] Hert L, Polymeris AA, Schaedelin S, Lieb J, Seiffge DJ, Traenka C, Fladt J, Thilemann S, Gensicke H, De Marchis GM, Bonati L, Lyrer P, Engelter ST, Peters N. Small vessel disease is associated with an unfavourable outcome in stroke patients on oral anticoagulation. Eur Stroke J. 2020 Mar;5(1):63-72. doi: 10.1177/2396987319888016. Epub 2019 Nov 12. PMID 32232171
- [Background] Cappellari M, Seiffge DJ, Koga M, Paciaroni M, Forlivesi S, Turcato G, Bovi P, Yoshimura S, Tanaka K, Shiozawa M, Yoshimoto T, Miwa K, Takagi M, Inoue M, Yamagami H, Caso V, Tsivgoulis G, Venti M, Acciarresi M, Alberti A, Toni D, Polymeris A, Bonetti B, Agnelli G, Toyoda K, Engelter ST, De Marchis GM; SAMURAI-NVAF, RAF-NOAC, NOACISP LONG-TERM, and Verona Study Groups. A nomogram to predict unfavourable outcome in patients receiving oral anticoagulants for atrial fibrillation after stroke. Eur Stroke J. 2020 Dec;5(4):384-393. doi: 10.1177/2396987320945840. Epub 2020 Nov 26. PMID 33598557
- [Background] Polymeris AA, Macha K, Paciaroni M, Wilson D, Koga M, Cappellari M, Schaedelin S, Zietz A, Peters N, Seiffge DJ, Haupenthal D, Gassmann L, De Marchis GM, Wang R, Gensicke H, Stoll S, Thilemann S, Avramiotis NS, Bonetti B, Tsivgoulis G, Ambler G, Alberti A, Yoshimura S, Brown MM, Shiozawa M, Lip GYH, Venti M, Acciarresi M, Tanaka K, Mosconi MG, Takagi M, Jager RH, Muir K, Inoue M, Schwab S, Bonati LH, Lyrer PA, Toyoda K, Caso V, Werring DJ, Kallmunzer B, Engelter ST; NOACISP-LONGTERM, Erlangen Registry, CROMIS-2, RAF, RAF-DOAC, SAMURAI-NVAF and Verona Registry Collaborators. Oral Anticoagulants in the Oldest Old with Recent Stroke and Atrial Fibrillation. Ann Neurol. 2022 Jan;91(1):78-88. doi: 10.1002/ana.26267. Epub 2021 Nov 29. PMID 34747514
- [Background] Seiffge DJ, Paciaroni M, Wilson D, Koga M, Macha K, Cappellari M, Schaedelin S, Shakeshaft C, Takagi M, Tsivgoulis G, Bonetti B, Kallmunzer B, Arihiro S, Alberti A, Polymeris AA, Ambler G, Yoshimura S, Venti M, Bonati LH, Muir KW, Yamagami H, Thilemann S, Altavilla R, Peters N, Inoue M, Bobinger T, Agnelli G, Brown MM, Sato S, Acciarresi M, Jager HR, Bovi P, Schwab S, Lyrer P, Caso V, Toyoda K, Werring DJ, Engelter ST, De Marchis GM; CROMIS-2, RAF, RAF-DOAC, SAMURAI, NOACISP LONGTERM, Erlangen and Verona registry collaborators. Direct oral anticoagulants versus vitamin K antagonists after recent ischemic stroke in patients with atrial fibrillation. Ann Neurol. 2019 Jun;85(6):823-834. doi: 10.1002/ana.25489. Epub 2019 Apr 30. PMID 30980560
- [Background] De Marchis GM, Seiffge DJ, Schaedelin S, Wilson D, Caso V, Acciarresi M, Tsivgoulis G, Koga M, Yoshimura S, Toyoda K, Cappellari M, Bonetti B, Macha K, Kallmunzer B, Cereda CW, Lyrer P, Bonati LH, Paciaroni M, Engelter ST, Werring DJ. Early versus late start of direct oral anticoagulants after acute ischaemic stroke linked to atrial fibrillation: an observational study and individual patient data pooled analysis. J Neurol Neurosurg Psychiatry. 2022 Feb;93(2):119-125. doi: 10.1136/jnnp-2021-327236. Epub 2021 Oct 11. PMID 34635567
- [Derived] Zietz A, Polymeris AA, Helfenstein F, Schaedelin S, Hert L, Wagner B, Seiffge DJ, Traenka C, Altersberger VL, Dittrich T, Kaufmann J, Ravanelli F, Fladt J, Fisch U, Thilemann S, De Marchis GM, Gensicke H, Bonati LH, Katan M, Fischer U, Lyrer P, Engelter ST, Peters N. The impact of competing stroke etiologies in patients with atrial fibrillation. Eur Stroke J. 2023 Sep;8(3):703-711. doi: 10.1177/23969873231185220. Epub 2023 Jul 4. PMID 37401394
- [Derived] Wagner B, Hert L, Polymeris AA, Schaedelin S, Lieb JM, Seiffge DJ, Traenka C, Thilemann S, Fladt J, Altersberger VL, Zietz A, Dittrich TD, Fisch U, Gensicke H, De Marchis GM, Bonati LH, Lyrer PA, Engelter ST, Peters N. Impact of type of oral anticoagulants in patients with cerebral microbleeds after atrial fibrillation-related ischemic stroke or TIA: Results of the NOACISP-LONGTERM registry. Front Neurol. 2022 Sep 20;13:964723. doi: 10.3389/fneur.2022.964723. eCollection 2022. PMID 36203998
- [Derived] Meya L, Polymeris AA, Schaedelin S, Schaub F, Altersberger VL, Traenka C, Thilemann S, Wagner B, Fladt J, Hert L, Yoshimura S, Koga M, Zietz A, Dittrich T, Fisch U, Toyoda K, Seiffge DJ, Peters N, De Marchis GM, Gensicke H, Bonati LH, Lyrer PA, Engelter ST. Oral Anticoagulants in Atrial Fibrillation Patients With Recent Stroke Who Are Dependent on the Daily Help of Others. Stroke. 2021 Nov;52(11):3472-3481. doi: 10.1161/STROKEAHA.120.033862. Epub 2021 Jul 27. PMID 34311567